CLINICAL TRIAL: NCT07383415
Title: Assessing the Effectiveness of Combined Intranasal Platelet-rich Plasma Plus Topical Insulin Versus Platelet-rich Plasma Alone in the Treatment of Post Inflammatory Anosmia: a Randomized Controlled Trial
Brief Title: Intranasal Platelet-Rich Plasma With or Without Topical Insulin for Post-Inflammatory Anosmia
Acronym: PRP-I RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amin Javer (Other)
Responsible Party: Sponsor-Investigator, Amin Javer, MD, St. Paul's Hospital, Canada
Organization: St. Paul's Hospital, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H25-02495
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Anosmia; Inflammatory Anosmia
Keywords: PRP; PRP-INSULIN
MeSH Terms: conditions — Anosmia | interventions — Insulin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP Plus Topical Insulin (Active Comparator): Participants receive intranasal platelet-rich plasma in combination with topical insulin.
  Interventions: Biological: Intranasal PRP Plus Topical Insulin
- PRP Alone (Placebo Comparator): Participants receive intranasal platelet-rich plasma with saline instead of insulin.
  Interventions: Biological: Intranasal PRP Plus Saline (Placebo)

INTERVENTIONS:
Biological: Intranasal PRP Plus Topical Insulin — Autologous platelet-rich plasma administered intranasally with the addition of topical insulin applied to the olfactory cleft.
  Arms: PRP Plus Topical Insulin
Biological: Intranasal PRP Plus Saline (Placebo) — Autologous platelet-rich plasma administered intranasally with saline applied in place of topical insulin as a placebo comparator.
  Arms: PRP Alone

SUMMARY:
This study evaluates whether adding topical insulin to intranasal platelet-rich plasma (PRP) improves smell recovery in adults with post-inflammatory anosmia. Participants will be randomly assigned to receive either intranasal PRP combined with topical insulin or intranasal PRP alone. Changes in olfactory function will be assessed over time to compare the effectiveness and safety of the two treatments.

DETAILED DESCRIPTION:
Post-inflammatory anosmia is a common cause of persistent olfactory dysfunction with limited effective treatment options. Platelet-rich plasma (PRP) has been proposed as a regenerative therapy due to its high concentration of growth factors, while topical insulin has demonstrated potential neurotrophic and anti-inflammatory effects in olfactory tissue.

This randomized controlled trial aims to evaluate whether the addition of topical insulin to intranasal PRP provides greater improvement in olfactory function compared with intranasal PRP alone in adults with post-inflammatory anosmia. Participants will be randomly assigned to receive either combined intranasal PRP plus topical insulin or intranasal PRP alone.

Olfactory function will be assessed at baseline and at predefined follow-up time points using validated smell testing methods. Safety and tolerability of the interventions will also be monitored throughout the study. The results of this study will contribute to understanding the potential role of regenerative and neurotrophic therapies in the management of post-inflammatory anosmia

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with olfactory dysfunction despite olfactory training therapy
* Loss of smell within the past 5 years
* Loss of smell occurred after an infection
* Platelet count is over 150,000 platelets per microliter

Exclusion Criteria:

Have a history of or currently have sinonasal tumours Have a history of surgery or radiotherapy for the base of your skull Have been treated with antibiotics in the past month before surgery Have a condition called systemic vasculitis or any bleeding disorder Have a suspected or known allergy to insulin or PRP or Platelet Lysate (PL) Have inhaled drugs (i.e cocaine) in the past 6 months of your enrollment Smell loss is due to a head trauma or after surgery Unable to complete the Sniffin Stick Smell test or questionnaires

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Olfactory Function | Baseline to 12 months post-intervention
  Change in olfactory function from baseline as measured using a validated smell identification test.

IPD SHARING:
Plan to Share IPD: Undecided